CLINICAL TRIAL: NCT02782793
Title: Predictors of Unsuccessful Endoscopic Mucosal Resection of Complex Colon Polyps: "You Can Look But You Can't Touch"
Brief Title: Predictors of Unsuccessful Endoscopic Mucosal Resection of Complex Colon Polyps
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: University of Colorado, Denver (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); University of California, Los Angeles (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Sri Komanduri, Director of Endoscopy, Northwestern University
Other Study IDs: STU00095441
Record Dates: First submitted 2016-05-12; First posted 2016-05-25 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Colon Polyps
Keywords: Endoscopic; Mucosal; Resection
MeSH Terms: conditions — Colonic Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient's with complex colon polyps
  Interventions: Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection

SUMMARY:
A prospective outcomes study in patients referred for endoscopic mucosal resection of complex colon polyps.

DETAILED DESCRIPTION:
Colon cancer is the third leading cause of cancer-related death in the United States. The number of these deaths has significantly decreased due to screening colonoscopies. A colonoscopy is a procedure in which a physician examines the rectum and large intestines for abnormalities through the use of a specialized camera called an endoscope. Colonoscopies decrease the mortality associated with colon cancer through two main ways: by detecting and removing pre-cancerous lesions called polyps; and by detecting colon cancer at earlier stage, when therapies can still be effective at treating or removing the cancer.

Most colon polyps are small and can be completely removed during a standard colonoscopy. However, there is a growing awareness amongst endoscopists of polyps that are too large or inaccessible to be safely removed during a routine colonoscopy. Previously, these lesions required surgery for removal of the affected part of the colon. There is a growing body of evidence that suggests these more complex colon polyps can be entirely removed endoscopically through a procedure called endoscopic mucosal resection (EMR), thereby avoiding costly and debilitating surgery. Given that it is a novel procedure, it is only available at specialized care centers.

EMR is a procedure identical to a colonoscopy, with more steps involved in the lifting and removal of complex polyps. As many as 80-90% of complex polyps can be successfully removed with EMR. However, it has been noted that removal of the polyp in pieces, rather than as a whole can result in a 20-30% recurrence rate at the resection site. Any manipulation of the polyp prior to EMR may impair the ability to fully remove the lesion. Some factors that have previously been suggested to increase the difficulty of EMR include previous dye injections, removal attempts, and polyp sampling. However, the true impact of previous manipulations of CCPs remains unclear.

This study aims to be one of the largest prospective, multi-centered studies investigating factors that predict the failure of EMR in the removal of complex colon polyps.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to each of the participating tertiary care centers for endoscopic mucosal resection (EMR)

Exclusion Criteria:

* Does not meet inclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Formation of a multi-site prospective database of patients refereed for endoscopic mucosal resection for a complex colon polyp(s).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Endoscopic and clinical factors which predict failure of resection of large colon polyps | 5 year follow up
  A systematic, prospective collection of data from a large cohorts of patients referred for colon EMR will provide useful data in effort to improve overall patient outcomes.

SECONDARY OUTCOMES:
Efficacy (%) of Endoscopic resection for large colon polyps | 5 year follow up
Factors which predict recurrence of adenoma after large polyp resection | 5 year follow up

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado, Denver, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No